CLINICAL TRIAL: NCT02326688
Title: Reliability of Kinematic Analysis in Assessment and Rehabilitation of the Upper Arm of Stroke Patients Following a Cerebral Vascular Accident, Hemiparetic Subjects
Brief Title: Quantification of Arm Non-Use After a Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 9368
Record Dates: First submitted 2014-12-15; First posted 2014-12-29 (Estimated); Last update posted 2014-12-29 (Estimated); Status verified 2014-12

CONDITIONS: Hemiplegia
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stroke patients (Experimental): Kinematic measurement of the amount of trunk displacement during a grasping task
  * Two separated measurements are recorded with a 6-hours interval
  * A third measurement provided by a second examinator is conducted
  Interventions: Other: Kinematic analysis of trunk compensation
- control patients (Experimental): Kinematic measurement of the amount of trunk displacement during a grasping task
  * Two separated measurements are recorded with a 6-hours interval
  * A third measurement provided by a second examinator is conducted
  Interventions: Other: Kinematic analysis of trunk compensation

INTERVENTIONS:
Other: Kinematic analysis of trunk compensation

SUMMARY:
Reproducibility assessment of a quantitative measure of the amount of trunk compensation by kinematic analysis in a grasping task in stroke patients.This "maladaptive trunk compensation" is suspected to be underlined by "arm non-use" in some patients, since this abnormal movement impairs the ability of patients to correctly flex their shoulder and extend their elbow during grasping.

ELIGIBILITY:
Inclusion Criteria:

* · Patient hemiparetic

  * Hemiplegic Patient
  * Patient can perform a global task with the gripping limb

Exclusion Criteria:

* Patient can not actively tender elbow of the affected limb,

  * Patient who can not actively flex the shoulder of the affected limb,
  * Patient with a passive extension deficit elbow> 30 °,
  * Patient with a shoulder flexion passive deficit> 60 °,
  * Patient with severe neglect
  * Patient bearer severe cognitive impairment
  * A patient with aphasia understanding disorders

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Kinematic measurement of trunk displacement by the maladaptive index trunk compensation | 1 day
  The Maladaptive Index Trunk Compensation (MTC) is the difference between the compensation index (CI) in the free trunk condition and to the fixed core condition. The compensation index is the core of the movement of the report on the movement of the hand.

CONTACTS AND LOCATIONS:
Locations (1):
- Uh Montpellier, Montpellier, France

REFERENCES:
- [Derived] Bakhti KKA, Laffont I, Muthalib M, Froger J, Mottet D. Kinect-based assessment of proximal arm non-use after a stroke. J Neuroeng Rehabil. 2018 Nov 14;15(1):104. doi: 10.1186/s12984-018-0451-2. PMID 30428896